CLINICAL TRIAL: NCT03835390
Title: SIMDiscovery: The Benefits of Utilizing a Preparation Program With Simulation in Reducing Anxiety and Increasing Preparedness Among Parents and Their Children Undergoing Spinal Fusion Surgery
Brief Title: SIMDiscovery: The Benefits of Utilizing a Simulation Preparation Program for Spinal Fusion Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Daniel Hedequist, Principle Investigator, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00030717
Record Dates: First submitted 2019-02-05; First posted 2019-02-08 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Scoliosis Idiopathic Adolescent
Keywords: Anxiety; Preparedness; Spinal Fusion
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants who agree to participate in the SIMDiscovery program will be asked if they would like to participate in the research. If they consent, they will fill out pre- and post-questionnaires concerning quality of life, anxiety levels concerning the surgery, and a knowledge assessment.
  Interventions: Behavioral: SIMDiscovery

INTERVENTIONS:
Behavioral: SIMDiscovery — The SIMDiscovery program consists of nine stations that were designed to mirror the different stages of the perioperative process. The stations mirror the different stages of the surgical process and provide patients and their families with education regarding what they can anticipate during each aspect of the intervention.

SUMMARY:
This is a pilot study aiming to examine preliminary effectiveness of a preparation program which includes simulation (SIMDiscovery) in reducing anxiety and increasing feelings of preparedness among parents and their children who will undergo spinal fusion surgery. SIMDiscovery is an experiential learning preparation program which aims to educate children and families about different medical procedures through simulation play.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents with adolescent idiopathic scoliosis and their parent(s)
* Spinal fusion surgery scheduled
* Developmental Age range (10+; no upper age range)
* Males and females of all races and ethnicities
* English-speaking families (although English need not be their primary language)
* Both patient and caregiver (when patient is under 18 years of age) are able to attend SIMDiscovery program

Exclusion Criteria:

* - Other significant chronic medical conditions (e.g., spina bifida, muscular dystrophy)
* Anterior surgical access
* ICU stay expected post-op
* Cognitive functioning level below 10yo

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Change from Parent's and Adolescent's Baseline Anxiety at 1 month using the State/Trait Anxiety Inventory | Baseline, 1 month
  Parent and adolescent anxiety will be measured at baseline utilizing the State/Trait Anxiety Inventory (STAI) (Spielberger et al., 1983). The STAI consists of 40 items total-20 items assessing trait anxiety (general proneness to anxious behavior) and 20 items assessing state anxiety (a current emotional state). All items are scored using a four-point scale (e.g., ranging from "Almost Never" to "Almost Always"). Scores can range from 20 to 80 with higher scores indicating greater anxiety. This measure has been validated for use with individuals ages 15 and above (Julian, 2011). If a patient is 15 years of age or above, they will complete the STAI, rather than the STAIC (see below).
Change from Child's Baseline Anxiety at 1 month using the State/Trait Anxiety Inventory for Children | Baseline, 1 month
  Child anxiety will be assessed utilizing the State/Trait Anxiety Inventory for Children (STAIC) (Spielberger & Edwards, 1973). Similar to the STAI, the STAIC consists of 20 items assessing state anxiety and 20 items assessing trait anxiety. Items are scored using a four-point scale and higher scores indicate greater anxiety. The STAIC has been validated for use with children up to age 15 years (Spielberger & Edwards, 1973).
Change from Parent's Baseline Feelings of Preparedness at 1 month using Caregiver Preparedness Scale | Baseline, 1 month
  Parent preparedness will be measured using the Caregiver Preparedness Scale (CPS) (Archbold, et al., 1990). This scale has been validated for use with adult caregivers (Petruzzo et al., 2017; Pucciarelli et al., 2014). The CPS includes eight items assessing caregiver preparedness to care for a patient's physical and emotional needs, setting up services, coping with the stress of caregiving, making caregiving activities pleasant for the caregiver and patient, responding and managing emergencies, obtaining assistance from the health care system, and overall preparedness. Each item is rated from 0 (not at all prepared) to 4 (Very well prepared). Items are summed for a total score that ranges from 0 to 32, with higher scores indicating feeling better prepared for the caregiving role.
Change from Child's Baseline Feelings of Preparedness at 1 month using a modified Caregiver Preparedness Scale | Baseline, 1 month
  In order to examine themes similar to parent preparedness but from the patient's perspective, we will administer a measure similar to the CPS (above) for children and adolescent patients. This measure has not been validated; rather, based on the validity of the CPS used to assess parent preparedness, we modified the measure to assess patients' perception of their ability to care for or advocate for themselves regarding their physical and emotional needs prior to the surgery. (Archbold, et al., 1990). All patients will complete this measure. This measure consists of six questions and similar to the CPS, each item is rated from 0 (not at all prepared) to 4 (Very well prepared). Items are summed for a total score that ranges from 0 to 24, with higher scores indicating more feelings of preparedness for the surgery.

SECONDARY OUTCOMES:
Knowledge of Perioperative Procedures measured by Spinal Fusion Knowledge Assessment | Baseline, 1 month
  Facts that patients learn through the preoperative appointment and the SIMDiscovery program measured by the Spine Fusion Knowledge Assessment developed by our team

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hedequist, MD, Principal Investigator — Boston Children's Hospital; Lauren Potthoff, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No